CLINICAL TRIAL: NCT03466931
Title: Efficacy of the "Milk Ladder" Intervention in the Development of Tolerance and the Recognition of B Cell Epitopes in Babies Who Are Allergic to Cow's Milk Proteins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Inmaculada Cerecedo, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Milk Ladder
Record Dates: First submitted 2018-02-02; First posted 2018-03-15 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: IgE-mediated Milk Allergy
MeSH Terms: interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention (Experimental): Meals containing Milk and Milk
  Interventions: Other: Milk
- Historical cohort (No Intervention): Standard care

INTERVENTIONS:
Other: Milk — Meals containing Milk and Milk
  Arms: Dietary intervention

SUMMARY:
Food allergies have become a relevant health problem in westernized societies, particularly, with children. Cow's milk (CM), along with hen's eggs, are the most common foods eliciting allergic reactions in children under 4 years of age. The main objective of this intervention study is to evaluate the safety and efficacy of the intervention known as "The Milk Ladder" in the development of tolerance by children with CM allergies. This will be compared to an historical cohort (CoALE), which investigated the natural history of this allergy. Additionally, the ability of informative epitopes will be evaluated for their potential to predict tolerance and their correlation against clinical variables.

The "Milk Ladder" will be evaluated within a prospective cohort of CM allergic children. This intervention is enacted through the introduction of meals cooked with progressively increasing amounts of cow's milk into the participant's diet. The primary outcome will be the development of tolerance which will be evaluated through a double-blind placebo-controlled food challenge. IgE and IgG4 epitopes will be described using a peptide microarray immunoassay. Quality of life will be determined by administering the FAQLQ-PF disease-specific questionnaire. Finally, within a subgroup of study participants, the ability of different peptides to activate basophils will be analyzed, and CM T cell epitopes will be studied by means of T-cell proliferation and cytokine production assays.

ELIGIBILITY:
Inclusion Criteria:

* Babies of both sexes.
* Age < 12 months.
* Clinical history of immediate reaction (<2 hours) after the intake of baby's formula and/or foods containing cow's milk.
* Sensitization to cow's milk proteins demonstrated by:

  * sIgE to cow's milk, alpha-Lactoabumin, beta-Lactoglobulin and/or Casein >0.1KU/l (ImmunoCAP®, ThemoFisher) and/or
  * Skin prick test to cow's milk, alpha-Lactoabumin, beta-Lactoglobulin and/or Casein ≥3mm
* If the reaction to milk occurred over 3 months before the recruitment, it will be mandatory to confirm reactivity to milk with an oral food test.
* Parents / legal representatives of the participant voluntary accept to participate.

Exclusion Criteria:

* Delayed reactions (> 2 h) after milk intake.
* Contact urticaria to milk if ingestion is well tolerated.
* Previous participation in oral tolerance induction/desensitization protocols.
* Treatment with any medication that might interfere the evaluation of the primary outcome or any study procedure.
* Any disease or condition which presents a contraindication to perform an oral challenge, either open or double-blind or any other study procedure.
* Social circumstances that might interfere with protocol adherence.
* Egg and/or wheat allergy (this exclusion criterion shall be verified before the beginning of the intervention).

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants that develop tolerance to milk after the 'Milk Ladder' intervention | 12 months
  Tolerance assessment: participants who successfully pass a double-blind placebo-controlled oral food challenge without experiencing any limiting symptom
Number of participants experiencing any adverse reaction | 12 months
  Number of participants experiencing any adverse reaction to milk-containing foods along the intervention assessed by Medical Dictionary for Regulatory Activities (MedDRA), version in place at the end of the study.
Change in antigen-specific IgE and IgG4 epitopes repertoire | 6 and 18 months
  Serum specific inmunnoglobulin levels using a milk peptide microarray immunoassay

SECONDARY OUTCOMES:
Quality of life | 6 and 18 months
  Change in quality of life total score during the intervention, assessed by the disease-specific questionnaire 'Food Allergy Quality of Life Questionnaire - Parent Form'
Potential T-cell epitopes | 12 months
  Identification of potential T-cell epitopes in serum assessed by a T lymphocyte proliferation assay and cytokine secretion
Ability of the milk allergenic peptides to activate basophils | 12 months
  In vitro determination of basophil activation upon antigen stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Cerecedo, e: MD, PhD, Study Chair — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided